CLINICAL TRIAL: NCT01813539
Title: A Phase I/II Study of ARGX-110 in Patients With Advanced Malignancies Expressing CD70.
Brief Title: A Study of ARGX-110 in Participants With Advanced Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OncoVerity, Inc. (Industry)
Collaborators: argenx (Industry); Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108755; ARGX-110-1201 (Other: Janssen Research & Development, LLC); 2012-005046-38 (EudraCT Number)
Record Dates: First submitted 2013-03-07; First posted 2013-03-19 (Estimated); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Neoplasms
Keywords: Malignancy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (10):
- Dose Escalation: Cohort 1 (Experimental): Participants will receive ARGX-110 as an intravenous infusion (IV) at dose level 1.
  Interventions: Drug: ARGX-110
- Dose Escalation: Cohort 2 (Experimental): Participants will receive ARGX-110 as an IV infusion at dose level 2.
  Interventions: Drug: ARGX-110
- Dose Escalation: Cohort 3 (Experimental): Participants will receive ARGX-110 as an IV infusion at dose level 3.
  Interventions: Drug: ARGX-110
- Dose Escalation: Cohort 4 (Experimental): Participants will receive ARGX-110 as an IV infusion at dose level 4.
  Interventions: Drug: ARGX-110
- Dose Escalation: Cohort 5 (Experimental): Participants will receive ARGX-110 as an IV infusion at intermediate dose level at the conclusion of Cohort 4 prior to opening the safety expansion cohorts to participants enrolment.
  Interventions: Drug: ARGX-110
- Safety Expansion: Cohort 1 (Experimental): Participants with solid tumors will receive ARGX-110 as an IV infusion at a dose based on the safety, PD, and PK profiles of ARGX-110 as per the dose escalation part of the trial.
  Interventions: Drug: ARGX-110
- Safety Expansion: Cohort 2 (Experimental): Participants with hematological malignancies (all etiologies) will receive ARGX-110 as an IV infusion at a dose based on the safety, PD, and PK profiles of ARGX-110 as per the dose escalation part of the trial.
  Interventions: Drug: ARGX-110
- Safety Expansion: Cohort 3 (Experimental): Participants with cutaneous T-cell lymphoma (CTCL) will receive ARGX-110 as an IV infusion at dose level 2 followed by a maintenance therapy at dose level 2 or 3.
  Interventions: Drug: ARGX-110
- Safety Expansion: Cohort 4 (Experimental): Participants with peripheral T-cell lymphoma (PTCL) will receive ARGX-110 as an IV infusion at dose level 2 followed by a maintenance therapy at dose level 2 or 3.
  Interventions: Drug: ARGX-110
- Exploratory Efficacy: Cohort 5 (Experimental): Participants with relapsed/refractory CTCL will receive ARGX-110 as an IV infusion followed by a maintenance therapy at dose level 3.
  Interventions: Drug: ARGX-110

INTERVENTIONS:
Drug: ARGX-110 — ARGX-110 will be administered as an IV infusion.

SUMMARY:
The purpose of this study is to determine the optimal dose of ARGX-110 in participants with advanced malignancies and to assess efficacy of ARGX-110 (exploratory efficacy cohort 5 only).

DETAILED DESCRIPTION:
Phase I study conducted in participants whose tumors express the target of interest. Pharmacokinetics (PK), pharmacodynamics (PD), biomarkers will be determined to support dose selection.

Phase II study conducted in Cutaneous T-cell lymphoma (CTCL) participants who are CD70 positive. PK, PD, biomarkers and immunohistochemistry (IHC) will be determined to assess efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of malignancy refractory to, or relapsing after standard therapy
* Solid tumors or T-cell malignancies positive for the CD70 antigen by Immunohistochemistry/Fluorescence-activated cell sorting (IHC/FACS) within 56 days prior to administering the first dose of ARGX-110. IHC criterion: greater than > 10 percent (%) of CD70 positive tumor cells
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, or 2
* Serum albumin greater than or equal to (>=) 20 gram per liter (g/L) (solid tumor only)
* Ability to comply with protocol-specified procedures/evaluations and scheduled visits. In particular, the ability of the patient to undergo a tumor biopsy (optional for safety expansion cohort 4)

Exclusion Criteria:

* History or clinical evidence of neoplastic central nervous system (CNS) involvement
* History of another primary malignancy that has not been in remission for at least 1 year
* Systemic glucocorticoid administration at doses greater than physiological replacement (prednisolone 20 milligram [mg] equivalent) within 28 days of ARGX-110 first dose administration (for T-cell malignancies higher systemic dose can be allowed following discussion with Sponsor)
* Major surgery within 28 days of ARGX-110 first dose administration
* Unresolved grade 3 or 4 toxicity from prior therapy, including experimental therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2013-02-27 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicity (DLT) | 21 days
  DLT is defined as drug-related grade 3 or 4 clinical adverse event (AE) occurring during the 21 days (3 weeks) following the first dose of ARGX-110.

SECONDARY OUTCOMES:
Plasma Concentrations of ARGX-110 | Up to 2 years
  Plasma concentration of ARGX-110 will be assessed.
Biomarkers (CD70 qPCR and sCD27) of ARGX-110 biological activity | Up to 2 years
  Biomarkers (CD70 quantitative polymerase chain reaction [CD70 qPCR] and soluble CD27 [sCD27]) will be measured in serum and on tumor samples to correlate systemic drug effects with AE and Tumor response.
Number of Participants who Achieve a Tumor Response | Up to 2 years
  Tumor response will be assessed according to RECIST.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (8):
- Belgium (3):
  - Brussels
  - Edegem
  - Ghent
- France (5):
  - Bordeaux
  - Lille
  - Paris
  - Pierre-Bénite
  - Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Silence K, Dreier T, Moshir M, Ulrichts P, Gabriels SM, Saunders M, Wajant H, Brouckaert P, Huyghe L, Van Hauwermeiren T, Thibault A, De Haard HJ. ARGX-110, a highly potent antibody targeting CD70, eliminates tumors via both enhanced ADCC and immune checkpoint blockade. MAbs. 2014 Mar-Apr;6(2):523-32. doi: 10.4161/mabs.27398. Epub 2013 Dec 6. PMID 24492296